CLINICAL TRIAL: NCT05418556
Title: Tailored Versus Coventional AntiPlaTelet Strategy Intended After OPTIMIZEd Drug
Brief Title: Tailored Versus Coventional AntiPlaTelet Strategy Intended After OPTIMIZEd Drug Eluting Stent
Acronym: OPTIMIZE-APT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Part of Cardiology, Principal Investigator, associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0568
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Intervention Model Description: * Eligible subjects will be randomized 1:1 to a) conventional DAPT strategy or b) tailored anti-platelet strategy (short DAPT followed by P2Y12 inhibitor alone) after optimized DES implantation guided by intravascular imaging.
  * All subjects will be clinically followed at 1, 6, and 12 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Arm (Active Comparator): After PCI, patients are prescribed aspirin at a daily dose of 100 mg PO plus a P2Y12 inhibitor [clopidogrel or ticagrelor or prasugrel according to the clinical diagnosis] for 12 months after the index PCI.
  Interventions: Drug: aspirin
- Tailored Arm (Experimental): The antiplatelet regimens post-PCI are 1-month DAPT (aspirin plus clopidogrel) followed by 11-months clopidogrel alone for CCS, and 3-months DAPT (aspirin plus P2Y12 inhibitor [ticagrelor, prasugrel]) followed by 9-months P2Y12 inhibitor alone for ACS.
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — DAPT strategy
  Other Names: clopidogrel; prasugrel; ticagrelor

SUMMARY:
Objectives: To assess the safety of tailored antiplatelet therapy (short DAPT followed by P2Y12 inhibitor alone strategy) in patients who received optimized DES implantation guided by intravascular imaging (IVUS or OCT)

Hypothesis: Tailored antiplatelet strategy (short DAPT followed by P2Y12 inhibitor alone) is superior to conventional antiplatelet strategy in terms of clinically relevant bleeding and noninferior for ischemic composite adverse events in patients who received intravascular imaging-guided optimized DES implantation. (Optimized stent evaluated by on-site IVUS/OCT could act as an essential criterion for decision making for tailored antithrombotic strategy)

DETAILED DESCRIPTION:
Objective: To assess the safety of tailored antiplatelet strategy (short DAPT followed by P2Y12 inhibitor alone) in patients who received optimized DES implantation guided by intravascular imaging (IVUS or OCT)

Design: Prospective, open label, multi-center, dual arm, randomized trial Number of Subjects 3,944 subjects (1972:1972) Study Population: Patients with coronary artery disease undergoing imaging-guided PCI

Study Design:

* Eligible subjects will be randomized 1:1 to a) conventional DAPT strategy or b) tailored anti-platelet strategy (short DAPT followed by P2Y12 inhibitor alone) after optimized DES implantation guided by intravascular imaging.
* All subjects will be clinically followed at 1, 6, and 12 months

Co-primary Endpoints:

1. Clinically relevant bleeding (BARC 2, 3, or 5) at 12 months post-PCI
2. Ischemic composite adverse events of all-cause death, MI, ischemia-driven TVR, stent thrombosis at 12 months post-PCI
3. Net clinical outcome (NACE) of all-cause death, MI, ischemia-driven TVR, stent thrombosis, BARC 2,3,5 bleeding at 12 months post-PCI

Statistics and Analysis: The study was designed to test the hypothesis that tailored antithrombotic strategy, as compared to the conventional DAPT, would be superior for clinically relevant bleeding, noninferior to the ischemic composite adverse events and NACE. The primary analysis would be evaluated by intention-to-treat analysis. With 3756 (each 1,878) patients, this study has >80% power to detect noninferiority of tailored antiplatelet strategy for ischemic composite adverse event, >85% power to detect noninferiority of tailored antiplatelet strategy for NACE, and >85% power to detect superiority of the tailored antiplatelet arm on clinically relevant bleeding. To compensate for 5% attrition rate, 3,944 (each 1,972) patients will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥19 years
2. Typical chest pain or objective evidence of myocardial ischemia suitable for PCI
3. Significant de novo coronary artery lesions suitable for DES implantation
4. Patients who underwent optimized stent implantation either by IVUS or OCT

   * Using IVUS

     * MSA >5.5 mm2, or MSA >90% of the MLA at the distal reference segment
     * Plaque burden <50% with 5 mm of both stent edge
     * No edge dissection, thrombus or plaque protrusion/stent area <10%
   * Using OCT

     * MSA >4.5 mm2, or MSA >90% of the MLA at the distal reference segment
     * No significant malapposition
     * No significant edge dissection, thrombus or plaque protrusion/stent area <10%
5. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

1. Angiographic exclusion criteria: any of the followings 1. Bypass graft lesions 2. Lesions in which impaired delivery of imaging catheters is expected:

   * Extreme angulation (≥90°) proximal to or within the target lesion.
   * Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   * Heavy calcification proximal to or within the target lesion.
2. In-stent restenosis
3. Hypersensitivity or contraindication to device material and its degradants and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated.
4. Persistent thrombocytopenia (platelet count <80,000/l)
5. Any history of hemorrhagic stroke or intracranial hemorrhage / TIA or ischemic stroke within the past 6 months
6. A known intolerance or hypersensitivity to a study drug (aspirin, clopidogrel or ticagrelor) or heparin
7. Patients requiring long-term oral anticoagulants or cilostazol
8. Any surgery requiring general anesthesia or discontinuation of aspirin and/or an ADP antagonist is planned within 12 months after the procedure.
9. A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
10. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
11. History of liver cirrhosis (Child-Pugh B or C) or biliary tract obstruction
12. Life expectancy < 1 years for any non-cardiac or cardiac causes
13. Cardiogenic shock at the index admission
14. Patient's pregnant or breast-feeding
15. Active bleeding or extreme-risk for major bleeding (e.g. active peptic ulcer disease, gastrointestinal pathology with a high risk for bleeding, malignancies with a high risk for bleeding)
16. Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3944 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1) clinically relevant bleeding [Bleeding Academic Research Consortium (BARC) 2, 3, or 5] | 12 month
  1) clinically relevant bleeding [Bleeding Academic Research Consortium (BARC) 2, 3, or 5]
2) net clinical outcome defined as a composite of all-cause death, MI, ischemia-driven target vessel revascularization (TVR), definite/probable stent thrombosis (ST), and clinically relevant bleeding [BARC 2, 3, or 5] | 12 month
  2) net clinical outcome defined as a composite of all-cause death, MI, ischemia-driven target vessel revascularization (TVR), definite/probable stent thrombosis (ST), and clinically relevant bleeding [BARC 2, 3, or 5]
3) ischemic composite adverse event of all-cause death, MI, ischemia-driven target vessel revascularization (TVR), definite/probable stent thrombosis (ST) | 12 month
  3) ischemic composite adverse event of all-cause death, MI, ischemia-driven target vessel revascularization (TVR), definite/probable stent thrombosis (ST)

SECONDARY OUTCOMES:
1) Major or minor bleeding according to definitions from TIMI and International Society of Thrombosis or Hemostasis (ISTH) | 12 month
  1) Major or minor bleeding according to definitions from TIMI and International Society of Thrombosis or Hemostasis (ISTH)
2) % difference of strut coverage on FU OCT between optimal vs. suboptimal DES implantation group | 1 or 3 month
  2) % difference of strut coverage on FU OCT between optimal vs. suboptimal DES implantation group

CONTACTS AND LOCATIONS:
Locations (25):
- South Korea (25):
  - Bucheon Sejong Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Chungbuk National University Hospital, Chungju
  - Daegu Catholic Univ Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Veterans Hospital, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Chungnam National University Sejong Hospital, Jungnam
  - Dankook University Hospital, Jungnam
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Veterans Hospital Service Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No